CLINICAL TRIAL: NCT06806345
Title: Effect of Hyperbaric Oxygen Therapy on Insulin Resistance in Postmenopausal Women
Brief Title: Hyperbaric Oxygen Therapy on Insulin Resistance in Postmenopause
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sherin Mohamed Samy Abdel Ghany Basha, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/004726
Record Dates: First submitted 2025-01-21; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Insulin Resistance Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Hyperbaric Oxygenation; Hypoglycemic Agents

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hyperbaric oxygen therapy group (Experimental): Hyperbaric Oxygen Therapy (HBOT): It was applied for Group (A) started with a gradual increase of oxygen pressure to be approximately 2.5 ATA through 15 min in a100% oxygen delivered for 60 min Then, gradual decompression through 15 min for a total of 90min per each session for 30 sessions (5 sessions per week for 6weeks)
  Interventions: Device: Hyperbaric oxygen therapy; Drug: Hypoglycemic Drug
- control group (Other): Hypoglycemic drug 'Metformin' Metformin reduces serum glucose level by several different mechanisms without increasing insulin secretion.it increases the effects of insulin so it is termed "insulin sensitizer ,metformin also suppresses the endogenous glucose production by the liver ,which is mainly due to a reduction in the rate of gluconeogenesis and asmall effect on glycogenolysis. Moreover, metformin activates the enzyme adenosine monophosphate kinase (AMPK) resulting in the inhibition of key enzymes involved in gluconeogenesis and glycogen synthesis in the liver while stimulating insulin signaling and glucose transport in muscles 500 mg once per day
  Interventions: Drug: Hypoglycemic Drug

INTERVENTIONS:
Device: Hyperbaric oxygen therapy — Hyperbaric Oxygen Therapy (HBOT):(Haux, Starmed 2300, Germany). A multichamper Double-lock, divided into Main chamber and Antichamber, with omega Ω-shape and all safety and CE-Certificate,
  Arms: hyperbaric oxygen therapy group
Drug: Hypoglycemic Drug — Metformin reduces serum glucose level by several different mechanisms without increasing insulin secretion.it increases the effects of insulin so it is termed "insulin sensitizer ,metformin also suppresses the endogenous glucose production by the liver ,which is mainly due to a reduction in the rate of gluconeogenesis and asmall effect on glycogenolysis. Moreover, metformin activates the enzyme adenosine monophosphate kinase (AMPK) resulting in the inhibition of key enzymes involved in gluconeogenesis and glycogen synthesis in the liver while stimulating insulin signaling and glucose transport in muscles

SUMMARY:
Background: In postmenopausal females, Insulin resistance is commonly encountered in clinical setting. Hyperbaric oxygen therapy have been proposed effective in lowering blood glucose level and improving function. Identification of clinical examination variables as predictors to blood glucose levels and dysfunction would offer therapists the chance to undertake clinical decisions and consequently improve treatment efficiency.

Objectives: This Predictive validity, diagnostic study conduct to examine the effect of hyperbaric oxygen therapy on insulin resistance in postmenopausal women.

DETAILED DESCRIPTION:
Purpose of the study:

The purpose of the current study is to determine if Hyperbaric oxygen therapy will have an effect on the treatment of post menopausal insulin resistance?

Significance of the study:

Insulin resistance along with Type2 diabetes (T2DM) is now considered an emerging clinical and public health problem in Egypt. Atherosclerotic cardiovascular diseases are the major causes of morbidity and mortality in diabetic patients (Soliman ,2008).

Persistent high glucose level leads to chronic damages and dysfunctions of various tissues, especially in the heart, blood vessel, eye, and kidney, causing a series of chronic complications. These complications(microvascular and macrovascular) are the major cause of disability in diabetic patients and has already been aserious social health. Thus, prevention and alleviation of the vascular complications has become a major challenge in diabetes therapy problem (Wang et al.,2015).

Hyperglycemia associated with diabetes mellitus causes vascular disease, which is responsible for most of the morbidity, hospitalizations, and death that occur in patients. Microvascular lesions promote nephropathy, retinopathy, and neuropathy, while damage to large blood vessels increase the risk of cardiovascular events by 2 to 4 folds(Buron and Thaunat,2020).

The goal of treatment for insulin resistance in postmenopausal women are to prevent or delay complications and maintain quality of life. This require control of glycemia, cardiovascular risk factor management,and regular follow-up. Life style modifications including physical activity , healthy diet ,smoking cessation and maintaince of ahealthy body weight are recommended as first line therapies from the time of diagnosis and as co-therapy for patients who also require glucose-lowering medications (Davies et al.,2018).

Hyperbaric oxygen therapy was found to improve glycemic control,increase insulin sensitivity in overweight or obese individuals with and without T2DM and improve atherogenic metabolic changes.suggested that it could be used as a therapeutic intervention for T2DM. ( Wilkinson et al.,2015)

ELIGIBILITY:
Inclusion Criteria:

* A)Inclusion Criteria

  * All females were clinically diagnosed with Postmenopausal Insulin resistance.
  * Their ages were ranged from 55-65 years old.
  * Their BMI was 30-34.9 kg/m².
  * All patients should had controlled blood glucose levels by oral hypoglycemic drugs.
  * All patients should had cardiac Ejection Fraction >or =50%.
  * Their Chest X-ray reported normal.
  * Their Ear ,nose , thorax will be clinically evaluated by a specialized ENT physician to ensure fitting for hyperbaric chamber
  * Voluntary acceptance of participation in the study .

B)Exclusion Criteria:

Participants will be excluded if they have :

* Chronic obstructive pulmonary disease.
* Cardiac pacemakers.
* Epileptic fits.
* Physically disable .
* Any disorder that lead to ulcers other than diabetes such as ahistory of chronic peripheral arterial disease.

Exclusion Criteria:

-

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal women
Enrollment: 40 (Estimated)
Dates: Start 2025-01-28 (Estimated); Primary Completion 2025-03-28 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
HgA1c | two months
  the glycated hemoglobin (HbA1c) level determines the ability of the body to control the glycemic level over the last 2-3 months, According to ADA, the HbA1C level for a normal subject is <5.7% and for adiabetic patient is >or=6.5%.
Function | two months
  Quality of life enjoyment satisfaction and questionnaire (QLES-QSFB):
  It consists of items that evaluate overall enjoyment and satisfaction regarding ; Physical Health, mood, work, household and leisure activities, family and social relationships, ability to function in daily life , economic status , living or housing situation , ability to get around physically, ability to do work or hobbies, and overall sense of being. The Q-LES-Q-SF is a validated, self reported evaluation of the degree to which enjoyment and satisfaction are derived from various areas of life . Responses were scored on a five point scale ( from "very poor" to " very good " ) , where higher scores indicate better enjoyment and satisfaction with life . Scores were added and presented as a percentage of the total maximum score . A percentage of total score of > 70 represents normal quality of life .
fasting blood glucose level | every 10 sessions for 2months
  The patients fasted for at least 8 hours. Measurements were done by blood glucose meter, a lancet device with lancets and test strips. The finger was picked with the lancet to obtain a very small drop of blood which was applied to a test strip placed in the meter.

CONTACTS AND LOCATIONS:
Locations (1):
- Kobry el koba military complex, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] 79, 1335-1340
- [Background] Golledge J, Singh TP. Systematic review and meta-analysis of clinical trials examining the effect of hyperbaric oxygen therapy in people with diabetes-related lower limb ulcers. Diabet Med. 2019 Jul;36(7):813-826. doi: 10.1111/dme.13975. Epub 2019 May 26. PMID 31002414
- [Background] Abildgaard J, Tingstedt J, Zhao Y, Hartling HJ, Pedersen AT, Lindegaard B, Dam Nielsen S. Increased systemic inflammation and altered distribution of T-cell subsets in postmenopausal women. PLoS One. 2020 Jun 23;15(6):e0235174. doi: 10.1371/journal.pone.0235174. eCollection 2020. PMID 32574226